CLINICAL TRIAL: NCT07202195
Title: Home-Based Neuromodulation Suits for Reducing Spasticity and Ataxia in Multiple Sclerosis: A Multi-center RCT
Brief Title: At Home Use of Stimulation Suits for Managing MS Symptoms
Acronym: HANDS-MS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Daphne Kos (Other)
Collaborators: Danish MS Hospitals, Haslev and Ry (Other); Universitair Ziekenhuis Brussel (Other); National MS Center Melsbroek (Other)
Responsible Party: Sponsor-Investigator, Daphne Kos, Professor, Universitair Ziekenhuis Brussel
Organization: Universitair Ziekenhuis Brussel (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: J5812540_2024
Record Dates: First submitted 2025-08-25; First posted 2025-10-01 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis; MS (Multiple Sclerosis); Spasticity With Multiple Sclerosis; Ataxia - Other; Ataxia, Cerebellar; Ataxia, Motor; Spasticity; Home Based Care
Keywords: ataxia; spasticity; multiple sclerosis; MS; neuromodulation suit; stimulation suit; exopluse molli suit; home-based rehabilitation; symptom management
MeSH Terms: conditions — Multiple Sclerosis; Cerebellar Ataxia; Ataxia; Muscle Spasticity | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stimulation suit group (Experimental): This group will wear a full-body stimulation suit every day or every other day for six weeks, in addition to their usual care.
  Interventions: Device: electro-stimulation suit; Other: Usual Care
- usual care (Other): This group will be a comparator and have no added intervention expect for their usual care.
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: electro-stimulation suit — In EXOPULSE Mollii Suit is a multi-channel full-body suit with a low energy electrical stimulation - 20 Volt and 20 Hz. It generates 2 milliamp pulses (into 0-10,000 Ohms) with the following parameters:
  * Pulse width: variable between 25 and 170 μs.
  * Length of period: 50 ms.
  * Maximum amplitude: 20 V. It is composed of a control unit, a jacket and pants, with 58 embed-ded electrodes, in direct contact with the skin, and pre-positioned to stimulate 40 key muscle groups.
  The suit comes in different sizes. A trained medical staff pre-programs which nerves/muscles to be stimulated based on a clinical assessment of the user and the outcome is evaluated through standardized methods. The stimulation program is thus specific to each user.
  Other Names: neuromodulation suit; stimulation suit; EXOPULSE MOLLII suit
  Arms: stimulation suit group
Other: Usual Care — The rehabilitation therapy that is being offered at the National MS Center Melsbroek, but somewhat reduced/adjusted to make time for initiation and follow-up of using the neuromodulation suit and potentially also during the weeks at home (i.e., rehabilitation being offered by municipalities).
  Other Names: standard care

SUMMARY:
This study is being carried out at Multiple Sclerosis (MS) centers to evaluate whether a full-body stimulation suit at home can help people with Multiple Sclerosis (pwMS) reduce symptoms like spasticity (muscle stiffness) and ataxia (poor coordination), and improve daily functioning.

Can pwMS who experience spasticity or ataxia benefit from using a stimulation suit for 6 weeks?

Researchers will compare two groups: an intervention group (who will use the suit) and a control group (who will not use the suit).

Participants in the intervention group will:

* Wear the suit for 6 weeks in total every day or every other day (1 week during their MS center admission and 5 weeks at home).
* Receive their usual care in addition to wearing the suit.
* Undergo clinical tests at the MS center after 1 week and 6 weeks of stimulation.

Participants in the control group will:

* Receive their usual care.
* Undergo clincial tests at the same time points as the other group.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants must have ataxia or spasticity alongside impairments in upper or lower extremity physical function. MAS score ≥ 1 will be used as an inclusion criterion to determine the presence of spasticity. SARA score ≥ 4 will be used as an inclusion criterion to determine the presence of ataxia. Note: one of the two criteria (MAS score or SARA score) must be fulfilled for a pwMS to be eligible.
* The patient must have the cognitive abilities to understand instructions and to be able to complete the questionnaires adequately
* Diagnosis of multiple sclerosis.

Exclusion Criteria:

* Implanted devices (like pacemaker, Baclofen pump, neurostimulator, defibrillator, shunts, ECG equipment, electronic life support, high frequency operation equipment )
* Change in disease modifying treatment within the last 3 months
* Use of Botuline Toxine A within the last 3months
* Recent relapse within the last 3 months
* Acute musculoskeletal problems that hinder the test performance,
* Pregnancy
* Sizes bigger than 3XL (triple eXtra Large)
* Skin eruptions and/or skin areas in the stimulation zone that are swollen, infected or inflamed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
NHPT+SSST score | After one and six weeks of stimulation for the intervention group. The control group will be assessed at the same time points.
  The primary outcome will be a combined measure of upper and lower extremity motor function, consisting of the Nine Hole Peg Test and the Six Spot step test (labelled NHPT+SSST score). Values are expressed in seconds.
  A higher score, indicates a worse outcome.

SECONDARY OUTCOMES:
Six spot step test (SSST) | SSST assessment will take place after weeks 1 and 6 of stimulation.
  Similar to the T25FW, the SSST is a quantitative measure of lower extremity function. The test contains a rectangular field with six circles on the floor following a criss-cross course. Five circles contain a block. The starting-point is the first circle, which does not contain a block. From there the patient walks to the other side of the field and kicks the blocks out of the five circles, as quickly as possible. The task is immediately administered again by having the patient walk back the same route. Both the dominant and non-dominant legs are tested twice.
  The Maximum value: 300.0 seconds A higher score indicates a worse outcome.
Nine Hole Peg Test (NHPT) | NHPT assessment will take place after weeks 1 and 6 of stimulation.
  The Nine-Hole Peg Test (NHPT) is an assessment tool used to evaluate movement speed, particularly fine hand motor skills. The patient must take nine pegs from a container as quickly as possible and place them into the holes on a board. Afterwards, the patient must remove the pegs and return them to the container. The time taken to complete the task is measured. The patient may only use the hand being tested and must repeat the procedure for each peg individually (they are not allowed to pick up multiple pegs at once).
  A higher score indicates a worse outcome.
Modified Ashworth Scale (MAS) | MAS assessment will take place during screening, as they are used to determine eligibility and after weeks 1 and 6 of stimulation.
  The Modified Ashworth Scale (MAS) is designed to objectively assess the degree of spasticity. The MAS measures the level of hypertonia in the left and right elbows and knees. The therapist evaluates the muscle tone and records the highest level of tone felt during five repetitions per joint, using a six-point scale (0 = no increase in muscle tone, 4 = limb rigid in flexion or extension and cannot be moved).
  A higher score indicates a worse outcome.
Scale for the Assessment and Rating of Ataxia (SARA) | SARA assessment will take place during screening, as they are used to determine eligibility and after weeks 1 and 6 of stimulation.
  SARA is a clinical scale which assesses a range of different impairments in cerebellar ataxia. The scale is made up of 8 items related to gait, stance, sitting, speech, finger-chase test, nose-finger test, fast alternating movements and heel-shin test.
  The minimum value: 0 The maximum value: 40 A higher score indicates a worse outcome.
Numeric Rating Scale (NRS) | NRS assessments will take place after weeks 1 and 6 of stimulation.
  The severity of ataxia and spasticity will be documented bij a numeric scale. The minimum value: 0 The maximum value: 10 A higher score indicates a worse outcome.
6 Minute walk test | The assessment will take place after weeks 1 and 6 of stimulation.
  The goal is for the participant to walk as many meters as possible within 6 minutes over a 30-meter course. The participant may use walking aids or foot orthoses. This test assesses the participant's functional capacity. The more meters walked, the better the functional capacity.
5 times sit to stand test (5STS) | The assessment will take place after weeks 1 and 6 of stimulation.
  De Timed Chair Stand Test is a simple evaluative test used to assess, among other things, muscle strength, balance, and fall risk in older adults. During the Timed Chair Stand Test, the patient is asked to stand up from a chair and sit down again five times as quickly as possible, without using the arms. The physiotherapist records the time in seconds. A score greater than 14s indicates a fall risk.
The patient-Determined Disease Steps (PDDS) | PDDS assessment will take place after weeks 1 and 6 of stimulation.
  A questionnaire on how a person with MS preceives their capacity to walk. The patient needs to chose one descrition the reflects their condition the best.
  The minimum value: 0 The maximum value: 8 A higher score, indicates a worse outcome.
The 12-item Multiple Sclerosis Walking Scale (MSWS12) | MSWS-12 assessment will take place after weeks 1 and 6 of stimulation.
  The 12-item Multiple Sclerosis Walking Scale (MSWS-12) is a self-report measure of the impact of MS on the individual's walking ability.
  The minimum value: 0 The maximum value: 100 A higher score, indicate a worse outcome.
The 36-item Manual Ability Measurement (MAM36) | MAM36 assessment will take place after weeks 1 and 6 of stimulation.
  The Manual Ability Measure (MAM) is designed as an outcome instrument to assess hand function based on the patient's responses to functional questions. Tasks are rated on a scale from 0 (cannot be done) to 4 (easy to do). Total scores range from 0 to 144.
  A higher score indicates greater perceived manual ability.
The EuroQol Questionnaire (EQ-D5) | EQ-5D assessment will take place after weeks 1 and 6 of stimulation.
  The EQ-5D is a standardized instrument that provides a score across five health dimensions: mobility, self-care, daily activities, pain/discomfort, and anxiety/depression. (5 items, three or five response categories) In addition, the patient must indicate how they perceive their overall health status on a scale from 0 to 100. To interpret the results correctly, it is important that the healthcare provider is familiar with the patient's demographic information. (8 items) A higher score indicates a worse outcome.
adapted Treatment Satisfaction Questionnaire for Medication version 1.4 (TSQM 1.4) | The adapted TSQM 1.4 assessment will take place after weeks 1 and 6 of stimulation. Only for the intervention group
  Is used to evaluate treatment satisfaction with the particular aim of development and evaluation of treatment satisfaction among the patients already undergoing treatment. TSQM (1.4) has 14 questions divided into 4 subscales: effectiveness (items 1 to 3), side effects (items 4 to 8), convenience (items 9 to 11), and global satisfaction (items 12 to 14). Higher scores indicate a higher patient satisfaction with medication (Liberato et al. 2020). The questions have been re-formulated so they are applicable to using the stimulation suit.
SymptoMScreen | SymptoMScreen assessment will take place weekly from the start of the intervention until end of the study.
  A tool for rapid assessment of MS symptom ( the six most common areas where symptomatic complaints occur and are discussed during clinical visits) severity in routine clinical practice. It uses a 7-point Likert scales for each functional domain (0 = not affected at all, 6 = total limitation/I'm unable to do most daily activities).
  The minimum value: 0 The maximum value: 72 A higher score indicates a worse outcome.
Modified Fatigue Impact Scales (MFIS) | The assessment will take place after weeks 1 and 6 of stimulation.
  The assessment will be used to assess the physical, cognitive, and psychosocial impact of fatigue. Each of the 21 items of the MFIS will be scored from 0-to-4, providing a total score ranging from 0 to 84 (higher scores, greater fatigue impact).

OTHER OUTCOMES:
Multiple Sclerosis (MS) type | Will be collected (at baseline) when a partcipant is found eligible
  MS type: primary progressive (PP), secundary progressive (SP), relapsing remitting (RR), ..
age | Will be collected at baseline when a partcipant is found eligible
  Age (years)
sex | Will be collected at baseline when a partcipant is found eligible
  sex (m/v)
height | Will be collected at baseline when a partcipant is found eligible
  height (cm)
weight | Will be collected at baseline when a partcipant is found eligible
  weight (kg),
Expanded Disability Status Score (EDSS) | Will be collected (at baseline) when a partcipant is found eligible
  latest EDSS: The Expanded Disability Status Scale measures your current level of disability.
  Values: (0.0 -10.0) A higher score indicates a worse outcome
Time since diagnosis | Will be collected (at baseline) when a partcipant is found eligible
  time since diagnosis (years)
Medication | Will be collected (at baseline) when a partcipant is found eligible
  Previous and current MS medication. previous and current ataxia or spasticity medication will be listed
Onset Spasticity and/or ataxia | Will be collected (at baseline) when a partcipant is found eligible
  Time since onset of ataxia or spasticity. (years)
Comorbidities | Will be collected (at baseline) when a partcipant is found eligible
  Comorbidities will be listed.

CONTACTS AND LOCATIONS:
Overall Officials: Daphne Kos, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (2):
- Nationaal MS Center Melsbroek, Steenokkerzeel, Belgium
- The Danish MS Hospitals, Ry, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weller LJR, Sherwood SM, Ng SH, Vellaichamy M, Noordin AA, Tan LY, Mahadev A, Yeo TH, Ng ZM. Can External Neuromodulation Garments Improve Gait and Function in Children With Cerebral Palsy? A Prospective Single-Arm Study. Health Sci Rep. 2025 Mar 23;8(3):e70566. doi: 10.1002/hsr2.70566. eCollection 2025 Mar. PMID 40129510
- [Background] Skjerbaek AG, Dalgas U, Stenager E, Boesen F, Hvid LG. The six spot step test is superior in detecting walking capacity impairments compared to short- and long-distance walk tests in persons with multiple sclerosis. Mult Scler J Exp Transl Clin. 2023 Dec 12;9(4):20552173231218127. doi: 10.1177/20552173231218127. eCollection 2023 Oct-Dec. PMID 38105806
- [Background] Riemenschneider M, Trenel P, Norgaard M, Boesen F. Multimethodological validation of the modified fatigue impact scale in a Danish population of people with Multiple Sclerosis. Mult Scler Relat Disord. 2022 Sep;65:104012. doi: 10.1016/j.msard.2022.104012. Epub 2022 Jul 2. PMID 35820358
- [Background] Rabin R, de Charro F. EQ-5D: a measure of health status from the EuroQol Group. Ann Med. 2001 Jul;33(5):337-43. doi: 10.3109/07853890109002087. PMID 11491192
- [Background] Perpetuini D, Russo EF, Cardone D, Palmieri R, De Giacomo A, Pellegrino R, Merla A, Calabro RS, Filoni S. Use and Effectiveness of Electrosuit in Neurological Disorders: A Systematic Review with Clinical Implications. Bioengineering (Basel). 2023 Jun 2;10(6):680. doi: 10.3390/bioengineering10060680. PMID 37370612
- [Background] Palmcrantz S, Pennati GV, Bergling H, Borg J. Feasibility and potential effects of using the electro-dress Mollii on spasticity and functioning in chronic stroke. J Neuroeng Rehabil. 2020 Aug 10;17(1):109. doi: 10.1186/s12984-020-00740-z. PMID 32778118
- [Background] Moller AB, Bibby BM, Skjerbaek AG, Jensen E, Sorensen H, Stenager E, Dalgas U. Validity and variability of the 5-repetition sit-to-stand test in patients with multiple sclerosis. Disabil Rehabil. 2012;34(26):2251-8. doi: 10.3109/09638288.2012.683479. Epub 2012 May 22. PMID 22612360
- [Background] Miller L, Mattison P, Paul L, Wood L. The effects of transcutaneous electrical nerve stimulation (TENS) on spasticity in multiple sclerosis. Mult Scler. 2007 May;13(4):527-33. doi: 10.1177/1352458506071509. Epub 2007 Jan 29. PMID 17463075
- [Background] Milinis K, Tennant A, Young CA; TONiC study group. Spasticity in multiple sclerosis: Associations with impairments and overall quality of life. Mult Scler Relat Disord. 2016 Jan;5:34-9. doi: 10.1016/j.msard.2015.10.007. Epub 2015 Oct 22. PMID 26856941
- [Background] McGinley MP, Goldschmidt CH, Rae-Grant AD. Diagnosis and Treatment of Multiple Sclerosis: A Review. JAMA. 2021 Feb 23;325(8):765-779. doi: 10.1001/jama.2020.26858. PMID 33620411
- [Background] Mai AS, Yong JH, Lim OZH, Tan EK. Non-invasive electrical stimulation in patients with neurodegenerative ataxia and spasticity: A systematic review and meta-analysis of randomized controlled trials. Eur J Neurol. 2022 Sep;29(9):2842-2850. doi: 10.1111/ene.15438. Epub 2022 Jun 27. PMID 35666142
- [Background] Learmonth YC, Motl RW, Sandroff BM, Pula JH, Cadavid D. Validation of patient determined disease steps (PDDS) scale scores in persons with multiple sclerosis. BMC Neurol. 2013 Apr 25;13:37. doi: 10.1186/1471-2377-13-37. PMID 23617555
- [Background] Jones AA, Purohit R, Bhatt T, Motl RW. Maintaining Mobility and Balance in Multiple Sclerosis: A Systematic Review Examining Potential Impact of Symptomatic Pharmacotherapy. CNS Drugs. 2025 Apr;39(4):361-382. doi: 10.1007/s40263-025-01159-7. Epub 2025 Feb 15. PMID 39954116
- [Background] Jakimovski D, Bittner S, Zivadinov R, Morrow SA, Benedict RH, Zipp F, Weinstock-Guttman B. Multiple sclerosis. Lancet. 2024 Jan 13;403(10422):183-202. doi: 10.1016/S0140-6736(23)01473-3. Epub 2023 Nov 7. PMID 37949093
- [Background] Hvid LG, Gaemelke T, Dalgas U, Slipsager MK, Rasmussen PV, Petersen T, Norgaard M, Skjerbaek AG, Boesen F. Personalised inpatient multidisciplinary rehabilitation elicits clinically relevant improvements in physical function in patients with multiple sclerosis - The Danish MS Hospitals Rehabilitation Study. Mult Scler J Exp Transl Clin. 2021 Feb 17;7(1):2055217321989384. doi: 10.1177/2055217321989384. eCollection 2021 Jan-Mar. PMID 33643662
- [Background] Hobart JC, Riazi A, Lamping DL, Fitzpatrick R, Thompson AJ. Measuring the impact of MS on walking ability: the 12-Item MS Walking Scale (MSWS-12). Neurology. 2003 Jan 14;60(1):31-6. doi: 10.1212/wnl.60.1.31. PMID 12525714
- [Background] Hahn A, Moeller S, Schlausch A, Ekmann M, de Chelle G, Westerlund M, Braatz F, Mayr W. Effects of a full-body electrostimulation garment application in a cohort of subjects with cerebral palsy, multiple sclerosis, and stroke on upper motor neuron syndrome symptoms. Biomed Tech (Berl). 2023 Sep 12;69(1):49-59. doi: 10.1515/bmt-2023-0271. Print 2024 Feb 26. PMID 38354212
- [Background] Gijbels D, Dalgas U, Romberg A, de Groot V, Bethoux F, Vaney C, Gebara B, Medina CS, Maamagi H, Rasova K, de Noordhout BM, Knuts K, Feys P. Which walking capacity tests to use in multiple sclerosis? A multicentre study providing the basis for a core set. Mult Scler. 2012 Mar;18(3):364-71. doi: 10.1177/1352458511420598. Epub 2011 Sep 27. PMID 21952098
- [Background] Feys P, Lamers I, Francis G, Benedict R, Phillips G, LaRocca N, Hudson LD, Rudick R; Multiple Sclerosis Outcome Assessments Consortium. The Nine-Hole Peg Test as a manual dexterity performance measure for multiple sclerosis. Mult Scler. 2017 Apr;23(5):711-720. doi: 10.1177/1352458517690824. Epub 2017 Feb 16. PMID 28206826
- [Background] Feys, P., Moghames, P., Kasilingam, E., King, R., Manacorda, T., Fonseca, M., Notas, K., & Kos, D. (2024). Prevalence, severity and impact of MS symptoms, and use of services in Europe: Results from the large scale IMSS survey. Multiple Sclerosis Journal, 30(3S), 1160.
- [Background] Cameron MH, Wagner JM. Gait abnormalities in multiple sclerosis: pathogenesis, evaluation, and advances in treatment. Curr Neurol Neurosci Rep. 2011 Oct;11(5):507-15. doi: 10.1007/s11910-011-0214-y. PMID 21779953
- [Background] Callesen J, Richter C, Kristensen C, Sunesen I, Naesby M, Dalgas U, Skjerbaek AG. Test-retest agreement and reliability of the Six Spot Step Test in persons with multiple sclerosis. Mult Scler. 2019 Feb;25(2):286-294. doi: 10.1177/1352458517745725. Epub 2017 Dec 20. PMID 29260609
- [Background] Buckley E, Mazza C, McNeill A. A systematic review of the gait characteristics associated with Cerebellar Ataxia. Gait Posture. 2018 Feb;60:154-163. doi: 10.1016/j.gaitpost.2017.11.024. Epub 2017 Dec 1. PMID 29220753
- [Background] Boesen F, Norgaard M, Trenel P, Rasmussen PV, Petersen T, Lovendahl B, Sorensen J. Longer term effectiveness of inpatient multidisciplinary rehabilitation on health-related quality of life in MS patients: a pragmatic randomized controlled trial - The Danish MS Hospitals Rehabilitation Study. Mult Scler. 2018 Mar;24(3):340-349. doi: 10.1177/1352458517735188. Epub 2017 Oct 6. PMID 28984159
- [Background] Bharmal M, Payne K, Atkinson MJ, Desrosiers MP, Morisky DE, Gemmen E. Validation of an abbreviated Treatment Satisfaction Questionnaire for Medication (TSQM-9) among patients on antihypertensive medications. Health Qual Life Outcomes. 2009 Apr 27;7:36. doi: 10.1186/1477-7525-7-36. PMID 19397800
- [Background] Amatya B, Khan F, Song K, Galea M. Effectiveness of Non-Pharmacological Interventions for Spasticity Management in Multiple Sclerosis: A Systematic Review. Ann Rehabil Med. 2024 Oct;48(5):305-343. doi: 10.5535/arm.240064. Epub 2024 Oct 31. PMID 39497494